CLINICAL TRIAL: NCT05579743
Title: Feasibility of Remote Wound Care: Implementing a Patient-Centered Remote Wound Monitoring Solution Using a Smartphone Application
Brief Title: Feasibility and Effectiveness of a Remote Monitoring Program for the Treatment of Diabetic Foot Ulcers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00292929; R03DK133557 (NIH)
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Foot; Diabetic Foot Ulcer; Wound; Foot; Wound Leg; Wound Heal; Diabetes Complications
MeSH Terms: conditions — Diabetic Foot; Foot Injuries; Diabetes Complications

STUDY DESIGN:
Intervention Model Description: Patients will be computer randomized 1:1 to receive wound care monitoring using remote diabetic foot ulcer (DFU) monitoring technology or standard in-person monitoring for 12 weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard care (No Intervention): Patients randomized to receive standard of care will be provided with a wound care plan at the time of enrollment, and then follow-up in clinic on a biweekly basis (week 2, 4, 6, 8, 10, 12) for a wound check and care plan update as needed.
- Remote wound monitoring technology (Experimental): Enrolled patients (and their caregivers, if applicable) are given an in-person training on how to use the smartphone app to self-assess their wound during regular dressing changes. Wound assessments are electronically transmitted to a secure, dedicated portal up to once a week for remote review by the study doctors. In-person follow-up is monthly (at the time of enrollment, week 4, week 8, and week 12).
  Interventions: Other: Remote wound monitoring technology

INTERVENTIONS:
Other: Remote wound monitoring technology — Healthy.io developed a professional-user wound management system that captures wound measurements and analyzes tissue distribution in real time through a smartphone application. Clinical oversight of the healing status of the wound via remote imaging and expert review allows for real time intervention when stagnation or worsening of a wound is detected. Patients with wounds on their legs will receive access to Healthy.io's mobile app and will be able to perform self-scans of their wound which will be automatically sent to the medical professionals, thus allowing them to assess the wound remotely.
  Arms: Remote wound monitoring technology

SUMMARY:
This research is being done to compare two different methods of wound monitoring for chronic wounds: remote wound monitoring using a smartphone app and in-person wound monitoring in a clinic setting. This will be a pilot non-blinded randomized controlled feasibility trial. The investigators will enroll 120 patients with an active diabetic foot ulcer (DFU) who present to the multidisciplinary diabetic foot clinic in Baltimore, Maryland. Patients will be computer randomized 1:1 to receive wound care monitoring using remote DFU monitoring technology or standard in-person monitoring for 12 weeks.

DETAILED DESCRIPTION:
The purpose of this research is to determine if a smartphone mobile application, also referred to as a mobile app or simply an app, designed to capture wound measurements and analyze wound tissue distribution in real-time, can be a practical patient-centered solution for regular wound management and assessment. The app will be compared to traditional in-person wound monitoring. One of the major limitations of most literature describing remote monitoring technologies is the lack of a control group. By randomizing half of the enrolled patients to remote monitoring via standard of care, the investigators will be able to compare patient and provider satisfaction with remote vs. in-person monitoring, as well as the wound healing outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged ≥ 18 years old
* In treatment for lower extremity wound related to diabetic foot ulcer
* Able and willing to use a smartphone to assess the wound for the duration of the study
* English language proficiency

Exclusion Criteria:

* Patients with less than 1 dressing change per week
* Patients with wound size that cannot be covered with a single app scan (out of boundary conditions include wounds that wrap around patient's entire leg)
* Patients with wounds in an inaccessible location who live without a caregiver to assist in taking wound scans

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-06 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who successfully complete a weekly wound scan | 12 weeks
  Overall weekly scan rate

CONTACTS AND LOCATIONS:
Overall Officials: Caitlin Hicks, MD, Principal Investigator — Johns Hopkins School of Medicine
Locations (1):
- Johns Hopkins University School of Medicine, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu YHA, Keegan AC, White MPS, Bose S, Leung SG, Sherman R, Abularrage CJ, Selvin E, Hicks CW. AI-Powered Remote Monitoring for Lower Extremity Wound Management: A Randomized Controlled Trial Protocol. JVS Vasc Insights. 2025 Aug 8:100279. doi: 10.1016/j.jvsvi.2025.100279. Online ahead of print. PMID 40857414